CLINICAL TRIAL: NCT05569993
Title: Does Glutamine Therapy Have a Positive Effect on Traumatic Brain Injury Patients?Double Blinded Randomized Clinical Trial
Brief Title: Glutamine and Traumatic Brain Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Engy Raafat Youssif, Assistant lecuturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Traumatic brain injury
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: 2 groups will recieve glutamine ,the other will be placcebo group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double blinded clinical trial Masking for patient,their relatives and outcome assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine group (Active Comparator): 30 patients will recieve .3 mg/kg of glutamine for first 7 days in ICU
  Interventions: Drug: Glutamine
- Placcebo group (Placebo Comparator): 30 patients will recieve placcebo for first 7 days in ICU
  Interventions: Other: Placcebo

INTERVENTIONS:
Drug: Glutamine — .3 mg/kg of glutamine
  Arms: Glutamine group
Other: Placcebo — Patients will recieve placcebo
  Arms: Placcebo group

SUMMARY:
Glutamate is an important neurotransmitter present in over 90% of all brain synapses and is a naturally occurring molecule that nerve cells use to send signals to other cells in the central nervous system.

Glutamate is a non-essential amino acid with restricted passage to the brain from the blood. In the CNS, glutamate is synthesised in neurons as part of the glutamate-glutamine cycle.5,6 so it plays an essential role in normal brain functioning and can improve situations related to impaired cognitive,motor and emotional functions and can be used to improve traumatic brain injury patient general health status

DETAILED DESCRIPTION:
The term "brain injury" covers a wide range of conditions and injuries relating to the brain, skull, and scalp. A traumatic brain injury (TBI) usually results when the head or body suffers from a violent blow or jolt that results in swelling, bruising, bleeding, or tearing of the brain tissue which any damage to it has the potential to change the way your body operates.

Now ,(TBI) is considered one of the major causes of disability and deaths ,As It contributes more than 30% Of deaths worldwide . Those who survive a TBI can face effects that last a few days, or the rest of their lives. Effects of TBI can include impaired motor, cognitive and emotional functioning. These issues not only affect individuals but can have lasting effects on families and communities.TBI can also cause some inflammatory mediators to be released in circulation that affect brain and systemic organs such as cortisol,IL6 and TNF etc. A lot of modialities have been introduced to help in decreasing these side effects.

Glutamine,a non-essential amino acid present abundantly throughout the body and is involved in many metabolic processes. It is synthesized from glutamic acid and ammonia. It is the principal carrier of nitrogen in the body and is an important energy source for many cells.glutamine has a restricted passage to the brain from blood but it is synthesised in the brain as a part of the glutamate-glutamine cycle.5,6 so it present in over 90% of all brain synapses and is a naturally occurring molecule that nerve cells use to send signals to other cells in the central nervous system,maintaining normal brain function and can improve situations related to impaired cognitive,motor and emotional functions.

Hypothesis of this study; Does glutamine therapy have a positive effect on traumatic brain injury patients ?

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old
* mild to moderate head trauma

Exclusion Criteria:

* patients with concurrent cns dysfunction
* Renal failure patient
* diabetic patients with neuropathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The duration of ICU stay | First 30 days
  The duration of ICU stay after glutamine adiminstration

SECONDARY OUTCOMES:
Consiousness level by Glagow coma scale | 30 days
  Glasgow coma scale improvement
The incidence of Convulsions | 30 days
  Convulsions controled by glutamine

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hassan Bakri, Professor, Study Chair — Assiut University; Emad Zarief Kamel, Assistant professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.google.com/url?sa=t&source=web&rct=j&url=https://www.mayoclinic.org/diseases-conditions/traumatic-brain-injury/symptoms-causes/syc-20378557&ved=2ahUKEwj03c7No736AhWJgP0HHWbdB_AQFnoECAsQAQ&usg=AOvVaw1hApNyp5Z15Rb6ZV9Bsz6j
- See also: Related Info — https://www.google.com/url?sa=t&source=web&rct=j&url=https://my.clevelandclinic.org/health/articles/22839-glutamate&ved=2ahUKEwj6lYmLpb36AhV0hv0HHXvCBlYQFnoECCsQAQ&usg=AOvVaw0I8zh85AIWxxVmICDoKYAD
- See also: https://www.google.com/url?sa=t&source=web&rct=j&url=https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4133642/&ved=2ahUKEwj6lYmLpb36AhV0hv0HHXvCBlYQFnoECEIQAQ&usg=AOvVaw1_kGwGwx5h2G2svqnAp1SJ — https://www.google.com/url?sa=t&source=web&rct=j&url=https://www.frontiersin.org/articles/10.3389/fnhum.2021.722323/full&ved=2ahUKEwj6lYmLpb36AhV0hv0HHXvCBlYQFnoECDAQAQ&usg=AOvVaw1Tp_hCCgkjNJLx_761AVQx
- See also: Related Info — https://www.google.com/url?sa=t&source=web&rct=j&url=https://medlineplus.gov/traumaticbraininjury.html&ved=2ahUKEwik8NOwpb36AhVUgP0HHZ9xDvQQFnoECEQQAQ&usg=AOvVaw1xT2gGMsCPiHuu0ZAFDDID